CLINICAL TRIAL: NCT02024906
Title: Effect of Soy Intake on Cardiovascular Disease Biomarkers in Subclinical Hypothyroid Participants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Jill Hamilton-Reeves, PhD RD LD (Other)
Collaborators: Soy Nutrition Institute (Unknown)
Responsible Party: Sponsor-Investigator, Jill Hamilton-Reeves, PhD RD LD, Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000073; UL1TR000001 (NIH); HD002528 (Other: Kansas Intellectual and Developmental Disabilities Research Center)
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Cardiovascular Disease; Subclinical Hypothyroid
Keywords: isoflavone; CVD; soy intake; subclinical hypothyroid
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Soybean Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- soy protein isolate (SPI) (Experimental): 25 grams soy protein isolate (SPI) containing approximately 30 mg/d isoflavones
  Interventions: Dietary Supplement: soy protein isolate (SPI)
- milk protein isolate (MPI) (Active Comparator): milk protein isolate (MPI) containing 0 mg/d isoflavones
  Interventions: Dietary Supplement: milk protein isolate (MPI)

INTERVENTIONS:
Dietary Supplement: soy protein isolate (SPI)
  Arms: soy protein isolate (SPI)
Dietary Supplement: milk protein isolate (MPI)
  Arms: milk protein isolate (MPI)

SUMMARY:
The purpose of this study is to help the researchers understand if using a soy supplement impacts cardiovascular disease risk factors in patients with subclinical hypothyroidism.

DETAILED DESCRIPTION:
This pilot trial is a double blind, randomized, parallel arm trial. Eighty participants with subclinical hypothyroidism will be randomized to consume either soy protein isolate or milk protein isolate for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with subclinical hypothyroidism (otherwise healthy volunteers)
* Adults aged 25 - 70 yrs.
* Willing to avoid consumption of soy/other isoflavone containing foods (i.e. some snack bars) during the study.
* Willing to avoid consumption of dietary (other than multivitamin) and herbal supplements during the study.

Exclusion Criteria:

* Taking drugs that interfere with thyroid function
* Planning pregnancy in the next 6 months
* Taking drugs that lower lipids, blood pressure, or sensitize insulin
* Regular consumption of soy products (>20 g/wk)
* Consumption of soyfoods within 90 days prior to enrollment.
* Known history of soy or milk allergy or intolerance.
* Taking antibiotics during the intervention
* Active viral infections such as Human immunodeficiency virus (HIV) positive or hepatitis

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes in the cardiometabolic profile | Change from Baseline to Week 8
  Evaluate the role of isoflavone intake on cardiovascular disease.

SECONDARY OUTCOMES:
Change in thyroid function | Change from Basesline to 8 Weeks
  Safety will be monitored through measuring thyroid stimulating hormone (TSH) and free thyroxine (T4) in participants while on the study.
Change in thyroid function | Change from Basesline to 4 Weeks
  Safety will be monitored through measuring thyroid stimulating hormone (TSH) and free thyroxine (T4) in participants while on the study.
Changes in the cardiometabolic profile | Change from Basesline to 4 Weeks
  Evaluate the role of isoflavone intake on cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Hamilton-Reeves, PhD, RD, LD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States